CLINICAL TRIAL: NCT04318210
Title: Open Label Extension (OLE) of the Study of the Safety and Efficacy of Daily Oral Antiretroviral Use for the Prevention of HIV Infection in Heterosexually Active Young Adults in Botswana
Brief Title: Open Label Extension (OLE) of the TDF2 Study, Botswana
Acronym: TDF2-OLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Botswana Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-4940-1
Record Dates: First submitted 2020-03-03; First posted 2020-03-23 (Actual); Results first posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: HIV Infections
Keywords: HIV incidence; HIV prevention; Tenofovir; Emtricitabine; Botswana; HIV seronegativity; PrEP
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TDF-FTC as PrEP (Experimental): Eligible HIV-uninfected participants were offered 12 months of oral Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg (TDF-FTC) once daily in the form of a single tablet regardless of their original study assignment in randomized phase.
  Interventions: Drug: Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg

INTERVENTIONS:
Drug: Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg
  Other Names: Truvada

SUMMARY:
This study is an open label and is an extension to the TDF2 study in which the investigators offered daily oral tenofovir/emtricitabine (TDF/FTC) for a maximum of 12 months to HIV uninfected former participants of the TDF2 study.

DETAILED DESCRIPTION:
This open label phase builds on a unique opportunity provided by the end of the randomized phase of the TDF 2 study. The randomized study provided a well-characterized cohort of persons who received standard prevention interventions, including monthly testing, counseling, and condoms. The primary intervention that will change in the open label phase is the provision of information about the demonstrated efficacy and safety of PrEP including counseling about how PrEP is not 100% effective, provision of open label rather than blinded study medication, and a shortened visit schedule designed to more closely approximate what would be feasible in an implementation program. This open label phase will therefore serve as an opportunity to gather additional information relevant to the delivery and uptake of daily oral PrEP that may help inform eventual more wide scale PrEP implementation in Botswana.The OLE also leverages unique opportunities to address important questions about how information about PrEP safety and efficacy might affect risk behavior. The randomized trial showed that condom use (81.9% in the TDF/FTC group and 79.7% in the placebo group, p = 0.21) and the number of participants with more than one sexual partner in the previous month (14.2% in the TDF/FTC group and 14.1% in the placebo group, p = 0.86) between the two groups was similar. The underlying premise of this OLE is that information about PrEP efficacy and the knowledge of taking active drug rather than placebo might alter perception of HIV risk. This extension seeks to determine whether this trend will occur in the cohort after individuals receive information and counseling about the partial protective efficacy of PrEP and to identify risk factors for changes in risk behavior. The randomized trial revealed that reported drug adherence between the two arms was almost identical at 84.1% in the TDF/FTC group and 83.7% in the placebo arm (p = 0.79). The investigators have designed this open label phase in order to determine 1) if the knowledge of receiving active drug and the receipt of information about PrEP safety and partial efficacy at the onset of the open label phase could have substantial effects on pill use and 2) to identify individual factors associated with this impact. In addition, the open label extension will provide more information about the long term safety of Truvada.

ELIGIBILITY:
Inclusion Criteria:

* Former TDF 2 participants
* Willing and able to provide informed written consent for participation
* If female, willing to use effective contraception during the trial (oral or injectable hormonal contraception, an intrauterine device [IUD], or who have had surgical interventions such as bilateral tubal ligation or hysterectomy)
* Laboratory values as follows within 30 days prior to enrollment:
* HIV uninfected by dual, parallel, rapid whole blood testing and HIV EIA
* Serum phosphorus ≥ 2.2 mg/dL
* Calculated creatinine clearance ≥ 60 mL/min

Exclusion Criteria:

* Positive urine pregnancy test (females)
* Breastfeeding (females)
* History of significant renal or bone disease
* Any other clinical condition or prior therapy that, in the opinion of the physician would make the subject unsuitable for the OLE or unable to comply with the dosing requirements

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 229 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Taylor, MD, MPH, Principal Investigator — Centers for Disease Control and Prevention

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared publicly without permission from the country of Botswana but may be available upon request.

RESULTS

PARTICIPANT FLOW:
Groups:
- TDF-FTC as PrEP: Eligible HIV-uninfected participants were offered 12 months of oral Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg (TDF-FTC) once daily in the form of a single tablet regardless of their original study assignment in randomized phase.
  Tenofovir Disoproxil Fumarate 300 mg + Emtricitabine 200 mg
Period: Overall Study
Arm/Group | TDF-FTC as PrEP
Started | 229
Completed | 153
Not Completed | 76

BASELINE CHARACTERISTICS:
Arm/Group | TDF-FTC as PrEP
Number analyzed (Participants) | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 229
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 30 [28 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 127
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 229
Region of Enrollment [Number; unit: participants]
  Botswana | 229
Enrollment Site [Count of Participants; unit: Participants]
  Gaborone | 132
  Francistown | 97
Education Level [Count of Participants; unit: Participants]
  Primary or less | 4
  Secondary | 141
  Post-secondary | 84
Marital Status [Count of Participants; unit: Participants]
  Single | 163
  Married | 18
  Cohabitating | 37
  Separated/Widowed | 11
Employment Status [Count of Participants; unit: Participants]
  Employed | 178
  Unemployed | 51
Had an HIV test since TDF2 Study [Count of Participants; unit: Participants]
  No | 17
  Yes | 212
Felt at risk for HIV [Count of Participants; unit: Participants]
  No | 46
  Yes | 183
Risk from partner for HIV [Count of Participants; unit: Participants]
  No | 73
  Yes | 156

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Drug Adherence Over the Past 3 Days
Description: A 30-day supply of TDF/FTC was dispensed at each monthly visit, for up to 12 months.
  Participants were asked monthly about their drug adherence and were asked to recall their time of dosing over the past 3 days.
  Question: "Please think back to [yesterday, 2 days ago, 3 days ago]. What time did you take Truvada? Was it in the morning, afternoon, evening, or you weren't able to take the pill that day?"
Time Frame: Up to 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | TDF-FTC as PrEP
Number analyzed (Participants) | 229
Participants
  Took daily dosage in past 3 days | 199
  Took 2 doses in past 3 days | 9
  Took 1 doses in past 3 days | 2
  No doses taken in past 3 days | 19

2. Primary Outcome: Number of Sex Partners
Description: Number of sex partners was assessed at baseline and each scheduled monthly visit, for up to 12 months.
  Responses to the following question refers to the number of partners reported in the past 30 days:
  "In the past 30 days, with how many partners have you had sexual intercourse?"
Time Frame: Up to 12 months
Population: Among 229 participants, 102 participants were women and 127 participants were men. Analyses were stratified by sex.
Measure: Mean (Standard Deviation); unit: sexual partners
Arm/Group | TDF-FTC as PrEP
Number analyzed (Participants) | 229
sexual partners
  Number of sex partners among women, overall: number analyzed (Participants) | 102
  Number of sex partners among women, overall | 0.87 (0.53)
  Number of sex partners among men, overall: number analyzed (Participants) | 127
  Number of sex partners among men, overall | 1.03 (0.74)

3. Primary Outcome: Number of Sex Acts by Condom Usage
Description: Number of sex acts by condom usage was assessed at baseline and each scheduled monthly visit, for up to 12 months.
  Responses to the following question refers to the number of sex acts with up to 3 partners.
  "In the past 30 days, how many times did you have sex with ['this partner']? When I ask about the number of times you had sex, please count each sexual act. For example, if you had 2 rounds of sexual intercourse with your partner on a single evening, count that as two times you had sex. Please remember that this only refers to vaginal and anal sex. It does not refer to oral sex."
  To assess condom use by sex act, the following question was asked to assess the number of sex acts with condoms and without condoms with up to 3 partners:
  "Of the ___ sex acts, how many times did you not use condoms the entire time?"
Time Frame: Up to 12 months
Population: Among 229 participants, 102 participants were women and 127 participants were men. Analyses were stratified by sex.
Measure: Mean (Standard Deviation); unit: sex acts
Arm/Group | TDF-FTC as PrEP
Number analyzed (Participants) | 229
sex acts
  Number of sex acts among women: number analyzed (Participants) | 102
  Number of sex acts among women | 4.01 (5.26)
  Number of sex acts among men: number analyzed (Participants) | 127
  Number of sex acts among men | 5.95 (6.67)
  Number of condomless sex acts among women: number analyzed (Participants) | 102
  Number of condomless sex acts among women | 1.28 (3.72)
  Number of condomless sex acts among men: number analyzed (Participants) | 127
  Number of condomless sex acts among men | 1.70 (4.34)
  Number of sex acts involving a condom among women: number analyzed (Participants) | 102
  Number of sex acts involving a condom among women | 2.72 (3.70)
  Number of sex acts involving a condom among men: number analyzed (Participants) | 127
  Number of sex acts involving a condom among men | 4.24 (5.19)

4. Primary Outcome: Extracellular Tenofovir (TFV) for Recent Drug Exposure
Description: Dried blood spots were collected at each monthly study visit to characterize drug adherence by measuring extracellular tenofovir (TFV) for recent drug exposure (~24 hours). Of 229 participants, 196 participants had monthly DBSs available for analysis. A sampling algorithm was designed to make inference to TFV and TFV-DP levels at all 12 months. For the TFV extracellular analysis, participants were randomly assigned to one of three sampling schedules, with equal probability: (a) months 1, 2, 5, 8, and 11; (b) months 1, 3, 6, 9, and 12; and (c) months 1, 4, 7, 10, and 12. These 196 participants contributed a total of 777 monthly DBSs for the TFV extracellular analysis.
  Extracellular TFV detectability was defined as having a mean TFV level (of up to four measurements) equal to or greater than 5 ng/mL.
Time Frame: Up to 12 months
Population: Of 229 participants, 196 participants had monthly DBSs available for analysis over a period of 12 months. These 196 participants contributed a total of 777 monthly DBSs for the TFV extracellular analysis.
Measure: Number; unit: number of DBS samples
Units Other Than Participants: Dried spot blood sample
Arm/Group | TDF-FTC as PrEP
Number analyzed (Participants) | 196
Number analyzed (Dried spot blood sample) | 777
number of DBS samples
  Detectable TFV | 713
  No detectable TFV | 64

5. Primary Outcome: Intracellular Tenofovir-diphosphate (TFV-DP)
Description: Dried blood spots were collected at each monthly study visit to characterize drug adherence by measuring intracellular tenofovir-diphosphate (TFV-DP) for long-term drug exposure (~7 days). The 196 participants who had monthly DBSs available were stratified by site, gender, and the 3 patterns previously assigned for the TFV extracellular analysis (2×2×3 = 12 strata). Then 60 participants were selected, 5 from each of the 12 strata, to balance by site, gender, and the above 3 patterns were maintained. In turn, the monthly DBSs indicated by the assigned pattern were analyzed. These 60 participants contributed a total of 237 monthly DBSs for the TFV-DP intracellular analysis. The observed TFV-DP levels in our study population were categorized as follows (units of drug in fmol/mL): 0 doses per week (<912); 1 dose taken per week (≥912 and <1824); 2 doses taken per week (≥1824 and <2688); 3 doses taken per week (≥2688 and <3600); 4 doses taken per week (≥3600 and <4464); 5 to 7 doses taken
Time Frame: Up to 12 months
Population: Of the 196 participants with monthly DBSs available over a period of 12 months, 60 participants were selected for TFV-DP intracellular analysis and contributed a total of 237 monthly DBSs for the TFV-DP intracellular analysis.
Measure: Number; unit: number of DBS samples
Units Other Than Participants: Dried blood spot sample
Arm/Group | TDF-FTC as PrEP
Number analyzed (Participants) | 60
Number analyzed (Dried blood spot sample) | 237
number of DBS samples
  7 doses per week | 141
  6 doses per week | 29
  5 doses per week | 20
  4 doses per week | 6
  3 doses per week | 12
  2 doses per week | 4
  1 dose per week | 5
  0 doses per week | 19

6. Secondary Outcome: HIV Seroconversion
Description: Study visits were scheduled every month until completion of the study and during monthly study visits, HIV testing was performed, for up to 12 months. During monthly visits, routine HIV testing was performed with two HIV rapid tests. If HIV-infection was suspected, HIV antigen-antibody (Ag/Ab) combination enzyme immunoassay (EIA) (Bio-Rad, GS HIV Combo Ag/Ab EIA) testing was performed, and RNA viral load was measured.
Time Frame: Up to 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | TDF-FTC as PrEP
Number analyzed (Participants) | 229
Participants | 0

7. Secondary Outcome: Serious Adverse Events
Description: Study visits were scheduled every month until study completion. Participants were instructed to return to the clinic for evaluation in event of illness. Participants reported any adverse effects (AEs) at monthly or interim visits and were determined as serious adverse events (SAE) when at least possibly related to study drug. DAIDS Table for Grading Severity of Adult Adverse Experiences for Vaccine & Prevention Research Programs was used for grading. Definitions: Grade 3-'probably related'-strong temporal relationship to study product that cannot be explained by participant's clinical state or other factors and a causal relationship is biologically plausible. Grade 4-'definitely related'-distinct temporal relationship to administration of the study product that cannot be explained by the participant's clinical state or other factors or AE occurs on re-challenge or the AE is a known reaction to the product or chemical group or can be predicted by the product's pharmacology.
Time Frame: Up to 12 Months
Measure: Number; unit: participants
Arm/Group | TDF-FTC as PrEP
Number analyzed (Participants) | 229
participants
  Hyperamylasemia, Grade 3 | 2
  Hypophosphatemia, Grade 3 | 5
  Hypercreatininemia, Grade 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the period of 12 months.
Arm/Group | TDF-FTC as PrEP
Serious Adverse Events (participants affected / at risk) | 8/229
Other Adverse Events (participants affected / at risk) | 169/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF-FTC as PrEP (N=229)
Hypophosphatemia (Blood and lymphatic system disorders) | 5 (6)
Hyperamylasemia (Blood and lymphatic system disorders) | 2 (2)
Elevated creatinine (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TDF-FTC as PrEP (N=229)
Hyperamylasemia (Blood and lymphatic system disorders) | 126 (223)
Hypophosphatemia (Blood and lymphatic system disorders) | 58 (89)
Transaminitis (Gastrointestinal disorders) | 22 (26)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 17 (23)
Headache (General disorders) | 21 (22)
Dizziness (Nervous system disorders) | 17 (22)
Hypocalcemia (Blood and lymphatic system disorders) | 15 (15)
Nausea (Gastrointestinal disorders) | 14 (14)
Vomiting (Gastrointestinal disorders) | 13 (13)
Pain, abdominal (Gastrointestinal disorders) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes